CLINICAL TRIAL: NCT02665338
Title: Repetitive TMS Modulates Dorsal Lateral Prefrontal-Ventral Medial Prefrontal Pathway to Decrease Craving in Smokers
Brief Title: TMS-fMRI for Neural Pathway in Smokers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We planned to enroll more participants but we could not recruit more participants. In addition, the covid-19 pandemic made the recruitment worse than the previous years.
Sponsor: Xingbao Li (Other)
Responsible Party: Sponsor-Investigator, Xingbao Li, Assistant Professor, Medical University of South Carolina
Organization: Medical University of South Carolina (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00032649
Record Dates: First submitted 2016-01-21; First posted 2016-01-27 (Estimated); Results first posted 2022-08-17 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-07

CONDITIONS: Nicotine Dependence
Keywords: transcranial magnetic stimulation; fMRI; cue craving
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Sham rTMS (Sham Comparator): The sham TMS system will be connected to an electrical generator on a 9 V battery and electrodes will be placed over the prefrontal cortex. The regulator is triggered by the TMS machine to allow brief, microsecond, pulses of the electrical current through to the skin on the subjects' forehead. Electrical stimulation will be triggered by the TMS machine to correspond to the sham TMS pulses.
  Interventions: Device: Transcranial Magnetic Stimulation
- Active rTMS (Active Comparator): Stimulation frequency for all active subjects: 10 Hertz - Pulse train duration (on time) 5 seconds, Inter-train interval (off time) 10 seconds (15 second cycle time), Power (intensity) level 100% rMT, Total 60 trains, 15 minutes, Total pulses 3000.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation
  Other Names: TMS

SUMMARY:
Cigarette smoking causes significant morbidity and mortality in the United States. Smoking cessation is difficult, with the average smoker attempting to quit five times before permanent success. Moreover, the majority of smoking quit attempts result in relapse. Brain stimulation for smoke cessation is an exciting new area that builds on advancing neuroscience knowledge concerning the functional neurocircuitry of addiction. Cortical stimulation can now be performed non-invasively by transcranial magnetic stimulation (TMS). Several studies have shown that TMS can reduce cue-elicited craving in smokers. Previous research by group has shown that a single session of 15 minutes high frequency (10 Hz) repetitive TMS (rTMS) at 100% motor threshold over the left dorsal lateral prefrontal cortex (DLPFC) can reduce cue-induced craving compared to sham TMS. However, the mechanism by which craving is reduced by rTMS is poorly understood both at behavioral and neural levels. Neuroimaging studies in nicotine dependence have revealed cue-related responses in numerous brain areas, including frontal, parietal cortices and subcortical areas. Recently functional magnetic resonance imaging (fMRI) studies by the group have shown that cue-induced craving induced brain activation in ventral medial prefrontal cortex (VMPFC), including medial frontal, orbital frontal and anterior cingulate. This Chair Research Development Fund (CRDF) pilot proposal will integrate two new techniques- TMS and fMRI to investigate DLPFC-VMPFC pathway in smokers. Using double-masked methods investigators hypothesize that cue-induced exposure will induce brain activity in VMPFC, and 15 minutes rTMS over DLPFC will reduce cue-induced craving through modulating DLPFC-VMPFC pathway (increased activity DLPFC and decreased activity VMPFC).

ELIGIBILITY:
Inclusion Criteria:

* Smoke 10 or more cigarettes per day and have a carbon monoxide (CO) level > 10 ppm indicative of recent smoking.
* Not received substance abuse treatment within the previous 30 days.
* Meet criteria for nicotine dependence as determined by the FTND.
* Be in stable mental and physical health.
* If female, test non-pregnant and use adequate birth control.
* No evidence of focal or diffuse brain lesion on MRI.
* Be willing to provide informed consent.
* Be able to comply with protocol requirements and likely to complete all study procedures.

Exclusion Criteria:

* Current dependence, defined by DSM-V criteria, on any psychoactive substances other than nicotine or caffeine.
* Contraindication to MRI (e.g., presence of metal in the skull, orbits or intracranial cavity, claustrophobia).
* Contraindication to rTMS (history of neurological disorder or seizure, increased intracranial pressure, brain surgery, or head trauma with loss of consciousness for > 15 minutes, implanted electronic device, metal in the head, or pregnancy).
* History of autoimmune, endocrine, viral, or vascular disorder affecting the brain.
* History or MRI evidence of neurological disorder that would lead to local or diffuse brain lesions or significant physical impairment.
* Unstable cardiac disease, uncontrolled hypertension, severe renal or liver insufficiency, or sleep apnea.
* Life time history of major Axis I disorders such as: Bipolar Affective disorder (BPAD), Schizophrenia, Post-traumatic Stress disorder (PTSD) or Dementia or Major Depression.
* Self report of >21 standard alcohol drinks per week in any week in the 30 days prior to screening.
* Other forms of nicotine delivery, such as nicotine patch, electronic cigarettes

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2014-04-28 (Actual); Primary Completion 2015-06-16 (Actual); Study Completion 2015-06-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Li X, Hartwell KJ, Owens M, Lematty T, Borckardt JJ, Hanlon CA, Brady KT, George MS. Repetitive transcranial magnetic stimulation of the dorsolateral prefrontal cortex reduces nicotine cue craving. Biol Psychiatry. 2013 Apr 15;73(8):714-20. doi: 10.1016/j.biopsych.2013.01.003. Epub 2013 Feb 26. PMID 23485014

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham rTMS: The sham TMS system will be connected to an electrical generator on a 9 V battery and electrodes will be placed over the prefrontal cortex. The regulator is triggered by the TMS machine to allow brief, microsecond, pulses of the electrical current through to the skin on the subjects' forehead. Electrical stimulation will be triggered by the TMS machine to correspond to the sham TMS pulses.
  Transcranial Magnetic Stimulation
- Active rTMS: Stimulation frequency for all active subjects: 10 Hertz - Pulse train duration (on time) 5 seconds, Inter-train interval (off time) 10 seconds (15 second cycle time), Power (intensity) level 100% rMT, Total 60 trains, 15 minutes, Total pulses 3000.
  Transcranial Magnetic Stimulation
Period: Overall Study
Arm/Group | Sham rTMS | Active rTMS
Started | 5 | 6
Completed | 5 | 5
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sham rTMS | Active rTMS | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Categorical [Count of Participants; unit: Participants] — Population: One subject did not complete all study.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 5 | 6 | 11
    >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (13.5) | 41.1 (13.4) | 39.7 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Changes in fMRI Neural Activation Patterns
Description: During MRI scan in which participants will watch smoking picture, investigators will measure the change in neural activity in reward neural circuit. Whole brain imaging analysis and network analysis will be performed.
Time Frame: 7 days
Population: Effect of rTMS on Cue-induced Brain Activity: Left accumbens and Right medial orbital frontal cortex.
Measure: Mean (Standard Error); unit: % change
Arm/Group | Sham rTMS | Active rTMS
Number analyzed (Participants) | 5 | 5
% change
  Left accumbens | 0.14 (0.09) | -0.38 (0.13)
  Right medial orbital frontal cortex | 0.13 (0.09) | -0.22 (0.1)

2. Secondary Outcome: Reduction of Smoking Cue Craving
Description: visual analog scale for cue craving. Participants will be asked ' Right now, I would rate the amount of my craving to smoke as:'. The minimum score is 0, and the Maximum score is 7. There are 10 items. The total minimum score is 0, and the total maximum score is 70. A higher score is more craving to smoke a cigarette. The fewer values are considered to be a better outcome.
Time Frame: pre-TMS and post-TMS approx, 30 minutes.
Population: The primary behavioral measure of cue craving was taken to be the contrast (difference) between active and sham rTMS in the pre- to post-experiment change in subjective craving. A two-factor mixed model (treatment: active vs sham) and (time: pre- vs post) were performed on cigarette-craving ratings.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sham rTMS | Active rTMS
Number analyzed (Participants) | 5 | 5
units on a scale
  Pre-TMS | 5.3 (2.4) | 6.8 (2.3)
  Post-TMS | 6.5 (2.1) | 6.4 (2.4)

ADVERSE EVENTS:
Time Frame: 7 days.
Description: During TMS treatment sessions, participants can feel pain, unpleasantness, or headache.
Arm/Group | Sham rTMS | Active rTMS
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham rTMS (N=5) | Active rTMS (N=6)
discomfort on head (Nervous system disorders) | 0 (0) | 1 (1) — The participant can feel discomfort in the head or headache.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes